CLINICAL TRIAL: NCT01249963
Title: Evaluation of Oral Enteral Nutrition Supplement in Patients With Mild Acute Pancreatitis
Brief Title: Enteral Nutrition Product in Mild Acute Pancreatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vegenat, S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: ATEM2010; Atémpero IDI-20080283 (Other: VEGENAT, S.A.)
Record Dates: First submitted 2010-11-26; First posted 2010-11-30 (Estimated); Last update posted 2012-06-22 (Estimated); Status verified 2011-02

CONDITIONS: Acute Pancreatitis; Enteral Nutrition
Keywords: acute pancreatitis; enteral nutrition; nutritional status; pancreas; T-Diet plus Atémpero
MeSH Terms: conditions — Pancreatitis | interventions — Phentermine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Group (Experimental): Patients of this group will receive 400 ml per day of T-Diet plus Atémpero product during 28 days.
  Interventions: Dietary Supplement: T-Diet plus Atémpero
- Control Diet (Active Comparator): Patients of this group will receive 2 packets (76 g) per day of AlitraQ (Abbott) product during 28 days.
  Interventions: Dietary Supplement: AlitraQ (Abbott)

INTERVENTIONS:
Dietary Supplement: T-Diet plus Atémpero — T-Diet plus Atémpero is a complete normocaloric and normoproteic enteral nutrition product for the dietary management of patients with mild acute pancreatitis.
  Other Names: ATEMP
  Arms: Experimental Group
Dietary Supplement: AlitraQ (Abbott) — AlitraQ is a nutritional product for patients with impaired gastrointestinal function.For oral or tube nutrition. Enriched with glutamine and arginine.
  Other Names: ALIT
  Arms: Control Diet

SUMMARY:
The aim of the study is to evaluate the beneficial effects of the administration of enteral nutrition product with milk proteins, monounsaturated fatty acids and low dextrose equivalent maltodextrin and enriched in eicosapentaenoic acid (EPA), docosahexaenoic acid (DHA) and medium chain triglycerides (MCT) in patients with mild acute pancreatitis. All this against other specific product.

The main objectives of this project are:

* Comparing the tolerance of both preparations.
* Comparing the evolution of nutritional status in both groups.
* Comparing the evolution of inflammatory parameters in both groups

DETAILED DESCRIPTION:
Oral administration of an oligomeric formula with milk proteins, mainly whey protein partially hydrolysate, monounsaturated fatty acids (AGM) and low dextrose equivalent maltodextrin and enriched in polyunsaturated fatty acids (PUFA) of omega-3 series, EPA and DHA, and MCT designed for nutritional support of patients with compromised intestinal function, to maintain or improve nutritional status and reduce the inflammatory response in undernourished patients with mild acute pancreatitis, compared with oligomeric enteral nutrition product, low in fat and rich in glutamine.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 with Mild Acute Pancreatitis.

Exclusion Criteria:

* Patients with Several Acute Pancreatitis
* Patients with life expectancy less than 48 hours.
* Renal (creatinin > 2,5 mg/dl) or kidney failure (GOT/GPT>2 from laboratory normal value)
* Patients with diabetes mellitus prior to acute pancreatitis.
* To take part in another study.
* Pregnant patients
* Informed consent absence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-02; Primary Completion 2012-12 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
Acceptance, Tolerance and Nutritional Status | 1 year
  * To compare the acceptance and tolerance of both products.
  * To compare the nutritional status in both arms.

SECONDARY OUTCOMES:
Inflammatory parameters evolution and EN complications | 1 year
  * To compare the inflammatory parameters evolution in both arms.
  * To evaluate the enteral nutrition complications.

CONTACTS AND LOCATIONS:
Overall Officials: Pilar García-Peris, PhD, Principal Investigator — Hospital Universitario Gregorio Marañón
Locations (1):
- Clinical Nutrition and Dietetic Unit, Hospital Universitario Gregorio Marañón, Madrid, Madrid, Spain